CLINICAL TRIAL: NCT06765707
Title: Symptom Monitoring Using Patient-Reported Outcomes to Optimize Medication Use
Brief Title: Symptom Monitoring Using Patient-Report to Improve Medication Use
Acronym: SyMPTOM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kathryn Flynn, Vice Chair, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRO00051010; 1R01CA285925-01A1 (NIH)
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3); Endocrine Therapy
Keywords: symptom management; symptom monitoring; pharmacist delivered intervention; oral endocrine therapy adherence
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Multi-center, two-arm cross-over, randomized control trial
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blinded for outcomes assessment for the 12-month outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care first, Then Symptom Monitoring and Management (Experimental): Patients first receive care as usual which includes follow-up with their oncology team first 12 months of the study. Following data collection at 12 months they will then receive symptom monitoring and management for the second 12 months of the study.
  Interventions: Behavioral: Pharmacist delivered symptom monitoring and management
- Symptom Monitoring and Management first, Then Usual Care (Experimental): Patients first receive symptom monitoring and management for the first 12 months of the study. After data collection at 12 months they will then receive care as usual which includes follow-up with their oncology for the second 12 months of the study.
  Interventions: Behavioral: Pharmacist delivered symptom monitoring and management

INTERVENTIONS:
Behavioral: Pharmacist delivered symptom monitoring and management — Patients in the intervention phase will receive PRO-based symptom monitoring once a month and pharmacist-led management for problematic symptoms based on routine clinical care recommendations.

SUMMARY:
This is an intervention targeting patients at risk for non-adherence to endocrine therapy after primary treatments for hormone-positive breast cancer. In a randomized study, the study team will collect patient-reported symptoms monthly from participants through surveys. Pharmacists who specialize in cancer at the patients' hospital will give patients recommendations to help improve their symptoms and address other barriers so they can continue daily endocrine therapy medications.

DETAILED DESCRIPTION:
This study will test whether oncology teams can adapt and combine models from intensive oncologic care and chronic noncancer care to support long-term oral oncologic medication adherence through better symptom monitoring and management. It will identify patients at risk of nonadherence through electronic health records and target them with a symptom monitoring and management intervention. The study will use patient-reported outcomes (PROs) to identify symptoms that may cause nonadherence and will involve clinical pharmacist-led follow-up.

Objectives:

1. Assess the impact of the intervention on adherence to oral endocrine therapy.
2. Evaluate the durability of adherence one-year post-intervention.
3. Describe the impact on symptoms and explore mechanisms for adherence improvement.

Intervention:

During the intervention phase, patients will receive symptom monitoring and pharmacist-led management based on patient-reported outcomes (PROs).

Symptom Monitoring:

1. Patients will report symptoms monthly for 12 months either online or via an interactive voice recording (IVR) system.
2. Symptoms will be assessed using PROs focusing on issues like pain, hot flashes, anxiety, and more.
3. Severe symptoms will trigger follow-up for management.

Symptom Management:

1. After the initial symptom report, patients will have a face-to-face or virtual visit with a clinical pharmacist.
2. The visit will be tailored based on patient preference and pharmacist judgment.
3. Pharmacists will discuss symptom reports, provide management recommendations, and coordinate with oncologists for prescriptions if needed.
4. All interactions will be documented in the electronic health record (EHR) for research analysis.

Control Phase:

Breast cancer patients on AET are typically seen every six months over a 5 to 10-year course, with more frequent visits if complications arise. Control group participants will continue to follow this schedule and receive an FDA document with tips for medication adherence.

Consent Process:

Informed consent will be obtained in person or remotely.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender women assigned female at birth
* Age 18 years or older
* Stage 1-3 hormone receptor-positive breast cancer

  1. Premenopausal patients being treated with GNRH agonist/antagonist to induce menopause are eligible
  2. Patients who received treatment with CDK 4/6 inhibitors are eligible
* Recommended to continue AET for ≥2 additional years after enrollment
* Low adherence defined as prescription fills with a proportion of days covered (PDC) of <80%, examined over all fills during the 2 years prior to date of eligibility review since the first AET prescription/data of AET start OR unable to calculate adherence
* Verbal fluency in English or Spanish
* Ability to understand informed consent and the willingness to sign it

Exclusion Criteria:

* Unable to verbalize comprehension of study or impaired decision-making
* Known distant metastatic disease
* Not receiving breast cancer care or AET prescription from provider at participating site
* Evidence that an oncology provider discontinued their AET
* Pregnant or trying to get pregnant
* Facility-administered medications (i.e., nursing home, home healthcare agency)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — People assigned female at birth who have not received masculinizing hormone therapy (that is, primarily cisgender women) will be included in this study. Although breast cancer occurs in cisgender men, trans women, and trans men, the use of endocrine therapy and its side effects can differ substantially across these groups particularly if they have previously received such therapy. Our intervention is structured around guideline concordant care based on research conducted in primarily cisgender women assigned female at birth, thus they are the primary focus at this stage. Nonbinary or transgender patients who were assigned female at birth and have not received hormone therapy would not, however, be excluded.
Enrollment: 225 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | From baseline to 12 months
  Defined as the proportion of total days' pills taken by patients measured by the opening of an electronic pill monitoring cap
Intervention durability on medication adherence | From 12 to 24 months
  Assess the durability of AET adherence 1 year post intervention on patients assigned to the intervention phase first. Defined as the proportion of total days' pills taken by patients measured by the opening of an electronic pill monitoring cap

SECONDARY OUTCOMES:
Medication adherence | From baseline to 12 months
  Medication adherence, based on prescription fill data (percent days covered, as used in screening)
Pain | From baseline to 24 months
  Patient-report collected via PROMIS Pain Interference measure
Fatigue | From baseline to 24 months
  Patient-report collected via PROMIS Fatigue measure
Sleep | From baseline to 24 months
  Patient-report collected via PROMIS Sleep-related Impairment measure
Anxiety | From baseline to 24 months
  Patient-report collected via PROMIS Anxiety measure
Depression | From baseline to 24 months
  Patient-report collected via PROMIS Depression measure
Sexual function | From baseline to 24 months
  Patient-report collected via PROMIS Sexual Function and Satisfaction measure
Physical functioning | From baseline to 24 months
  Patient-report collected via PROMIS Physical Functioning measure.
Social functioning | From baseline to 24 months
  Patient-report collected via PROMIS Ability to Participate in Social Roles and Activities measure
Self-efficacy to manage medications | From baseline to 24 months
  Patient-report collected via PROMIS Self-efficacy to Manage Medications measure
Self-efficacy to manage symptoms | From baseline to 24 months
  Patient-report collected via PROMIS Self-efficacy to Manage Symptoms measure
Social support | From baseline to 24 months
  Patient-reported collected via PROMIS Instrumental Support measure
Team-patient communication quality | From baseline to 12 months
  Team-patient communication quality collected using The Communication Assessment Tool

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Illinois Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
For patients who consent to sharing, the cleaned, de-identified, individual-participant level scientific data for all variables used in the analyses that address the specific aims will be shared, along with example transformations from initial raw data.
Supporting Information: Study Protocol
Time Frame: Shared data generated from this project will be made available no later than 12 months after the funding period ends. The duration of preservation and sharing of the data will be a minimum of 10 years after the funding period.
Access Criteria: There are no anticipated factors or limitations that will affect the access, distribution or reuse of the de- identified scientific data generated by the proposal. The de-identified scientific data that is shared will be shared by unrestricted download via Harvard Dataverse.

REFERENCES:
- [Background] Neuner J, Weil E, Fergestrom N, Stolley M, Kamaraju S, Oxencis C, Winn A, Laud PW, Flynn KE. Feasibility of a pharmacist-led symptom monitoring and management intervention to improve breast cancer endocrine therapy adherence. J Am Pharm Assoc (2003). 2022 Jul-Aug;62(4):1321-1328.e3. doi: 10.1016/j.japh.2022.03.001. Epub 2022 Mar 5. PMID 35393248